CLINICAL TRIAL: NCT01804816
Title: Acupuncture on Cardiac and Autonomic Function in Human Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wilson Tang, Staff Cellular and Molecular Medicine and Cardiovascular Medicine, The Cleveland Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 12-580
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Acupuncture (Experimental): 10 standardized verum acupuncture (VA) sessions twice a week, over 5 weeks. The 5 weeks of acupuncture were scheduled after the period of no acupuncture for each subject.
  Interventions: Procedure: Acupuncture
- No Acupuncture (Placebo Comparator): No acupuncture treatment or other study intervention over 5 weeks. All subjects had a 5 week period of "no acupuncture" prior to the 5 weeks of acupuncture sessions.
  Interventions: Other: No Intervention

INTERVENTIONS:
Procedure: Acupuncture — Standardized acupuncture administration for 10 sessions.
  Arms: Acupuncture
Other: No Intervention — No intervention during this period. This was a control period. Each subject acted as their own control.
  Arms: No Acupuncture

SUMMARY:
Acupuncture treatment may improve the cardiac function and the quality of life in heart failure patients. These effects may be related to the inhibition of sympathetic activity and/or increased vagal function. The suppression of inflammatory reaction with acupuncture treatment may also be associated with these outcomes. Specific aims include:

1. To evaluate the effect of acupuncture treatment on human cardiac sympathetic/vagal activity
2. To evaluate the effect of acupuncture treatment on cardiac function and functional capacity
3. To evaluate the general health score of the quality-of-life with acupuncture treatment
4. To explore the mechanism of acupuncture treatment on inflammation and nitrative stress in heart failure patients.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the effect of acupuncture treatment on cardiac sympathetic/vagal activity in chronic heart failure patients. The investigators would like to investigate the effect of acupuncture treatment on cardiac function and the general health score of the quality-of-life. The investigators would like to further explore the mechanism of acupuncture treatment on autonomic imbalance and chronic inflammatory reaction in heart failure patients by comparing the treatment and sham groups, the baseline before the treatment and the changes after treatment.

Chronic heart failure affects millions people and is a leading cause of death in US. Despite of advance in diagnoses and treatments, the long-term prognosis and quality of life of chronic heart failure patients remain poor. The mortality of chronic heart failure is estimated 50% within 4 years, and is more than 50% in patients with severe chronic heart failure.

Chronic heart failure results from the left ventricular (LV) systolic and/or diastolic dysfunction. Autonomic imbalance with sustained sympathetic overdrive and vagal withdrawal plays an important role in the development of chronic heart failure. This autonomic dysregulation is related to increased heart rate, excess inflammatory response, progressive LV dysfunction, increased mortality and morbidity in chronic heart failure patients. Sympathetic active inhibition with beta-adrenergic receptor blockers has shown significant reduction in mortality and morbidity in chronic heart failure patients. Also modulation of parasympathetic activation with electrical vagus nerve stimulation (VNS) has demonstrated as a potential therapy for chronic heart failure.

Acupuncture has been widely used in China for thousands of years to treat a variety of diseases and their symptoms. Except pain disorders, increasing evidences have shown that acupuncture may be useful for cardiovascular diseases, such as coronary artery disease, hypertension and chronic heart failure. It has been demonstrated that certain acupuncture points have shown to inhibit cardiac sympathetic activation or increase cardiac vagal component in both experimental animals and clinical studies. Recently a small clinical trial by Dr. Kristen, et al has found that acupuncture could improve exercise tolerance in chronic heart failure patients.

The investigators hypothesize that acupuncture treatment may improve the cardiac function and the quality of life in heart failure patients. These effects may be related to the inhibition of sympathetic activity and/or increased vagal function. The suppression of inflammatory reaction with acupuncture treatment may also be associated with these outcomes. In addition to optimized standard heart failure medications, acupuncture may be a safe therapeutic strategy in chronic heart failure treatment. Studies of acupuncture on cardiac autonomic activity in heart failure may show more evidence of acupuncture treatment in chronic heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Congestive Heart Failure (CHF), New York Heart Association (NYHA) class II-III, Left Ventricular Eject Fraction (LVEF) ≤40%
* All patients will have sinus rhythm and compensate with individually optimized standard heart failure medications. Routine medications will be continued during the study period
* Able and willing to give informed consent or comply with study procedures.

Exclusion Criteria:

* Acupuncture treatment within 3 months before the beginning of the study
* Presents with cutaneous eczema at potential acupoints
* Have a history of major bleeding or increased propensity of excessive bleeding due to platelet dysfunction
* Currently taking anti-coagulants (e.g. warfarin)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2015-01-09 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W.H. Wilson Tang, MD, Principal Investigator — The Cleveland Clinic; Yanming Huang, MD PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual patient data available.

REFERENCES:
- [Background] Middlekauff HR, Hui K, Yu JL, Hamilton MA, Fonarow GC, Moriguchi J, Maclellan WR, Hage A. Acupuncture inhibits sympathetic activation during mental stress in advanced heart failure patients. J Card Fail. 2002 Dec;8(6):399-406. doi: 10.1054/jcaf.2002.129656. PMID 12528093
- [Background] Kurono Y, Minagawa M, Ishigami T, Yamada A, Kakamu T, Hayano J. Acupuncture to Danzhong but not to Zhongting increases the cardiac vagal component of heart rate variability. Auton Neurosci. 2011 Apr 26;161(1-2):116-20. doi: 10.1016/j.autneu.2010.12.003. Epub 2011 Jan 7. PMID 21216208
- [Background] Deng YJ, Liang WX, Cheng SY. [Influence of acupoint-catgut-implantation on blood pressure and cardiac function in chronic congestive heart failure rats]. Zhen Ci Yan Jiu. 2011 Feb;36(1):40-5. Chinese. PMID 21585058
- [Background] Kristen AV, Schuhmacher B, Strych K, Lossnitzer D, Friederich HC, Hilbel T, Haass M, Katus HA, Schneider A, Streitberger KM, Backs J. Acupuncture improves exercise tolerance of patients with heart failure: a placebo-controlled pilot study. Heart. 2010 Sep;96(17):1396-400. doi: 10.1136/hrt.2009.187930. Epub 2010 Jun 15. PMID 20554511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Cleveland Clinic Heart and Vascular Institute section of Heart Failure and Transplant Medicine.
Pre-assignment Details: All subjects acted as their own controls for this study and were assigned to a 5 week period of no acupuncture or other study interventions (control) followed by a 5 week period of weekly standardized verum acupuncture (intervention).
Groups:
- No Acupuncture / Acupuncture: 5 weeks of no treatment followed by 5 weeks of standardized verum acupuncture.
Period: No acupuncture (initial 5 weeks)
Arm/Group | No Acupuncture / Acupuncture
Started | 14
Completed (Completed all study procedures.) | 11
Not Completed | 3
Not completed — Withdrawal by Subject | 3
Period: Acupuncture (second 5 weeks)
Arm/Group | No Acupuncture / Acupuncture
Started | 11
Completed | 10
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- No Acupuncture/Acupuncture: No Acupuncture: No treatment. Baseline period. Acupuncture: Standardized acupuncture administration for 10 sessions using acupuncture needles.
Arm/Group | No Acupuncture/Acupuncture
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Cardiac Function: LVEF
Description: Left ventricular ejection fraction (LVEF) percentage was measured at baseline, after 5 weeks of no treatment and just prior to acupuncture treatment, and after 5 weeks of acupuncture treatments.
Time Frame: Baseline, Week 7, Week 13
Measure: Mean (Standard Deviation); unit: LVEF Percentage
Groups:
- Baseline: Measurements at baseline visit.
- Pre-Acupuncture: Measurements were taken after 5 full weeks of no treatment. This visit occurred 6-7 weeks after the baseline measurements.
- Post-Acupuncture: Measurements were taken after 10 sessions of standardized verum acupuncture administration using 0.18-0.25×30-60-mm stainless steel needles. Acupuncture sessions were scheduled twice a week for 5 weeks. This post-acupuncture visit occurred within 1 week of finishing the acupuncture sessions.
Arm/Group | Baseline | Pre-Acupuncture | Post-Acupuncture
Number analyzed (Participants) | 10 | 10 | 10
LVEF Percentage | 36.14 (7.23) | 36.11 (8.97) | 40.59 (9.28)
Statistical Analysis 1: Comparison: Baseline vs Post-Acupuncture; Test type: Equivalence — a=0.05; p = 0.063, t-test, 2 sided

2. Primary Outcome: Change in 6-Minute Walk Distance
Time Frame: Baseline, Week 7, Week 13
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Baseline | Pre-Acupuncture | Post-Acupuncture
Number analyzed (Participants) | 10 | 10 | 10
Feet | 1376.2 (250.19) | 1488.0 (264.82) | 1515.10 (268.98)
Statistical Analysis 1: Comparison: Baseline vs Pre-Acupuncture; Based on results from prior small clinical trials we estimate the need for 20 patients enrolled to reach 80% statistical power; Test type: Equivalence — a = 0.05; p = 0.005, t-test, 2 sided
Statistical Analysis 2: Comparison: Baseline vs Post-Acupuncture; Test type: Equivalence — a=0.05; p = 0.002, t-test, 2 sided
Statistical Analysis 3: Comparison: Pre-Acupuncture vs Post-Acupuncture; Test type: Equivalence — a=0.05; p = 0.441, t-test, 2 sided

3. Secondary Outcome: Change in Quality of Life (QOL)
Description: Patients quality of life (QOL) was assessed using the Kansas City Cardiomyopathy Questionnaire (KCCQ) at baseline, after 5 weeks of no treatment and just prior to acupuncture treatment, and after 5 weeks of acupuncture treatments. Scores reported here are the Quality of Life Scores, which range from 0 to 100. Higher numbers indicate a better quality of life.
Time Frame: Baseline, Week 7, Week 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Pre-Acupuncture | Post-Acupuncture
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 65.00 (26.59) | 67.50 (24.36) | 69.17 (25.78)
Statistical Analysis 1: Comparison: Baseline vs Post-Acupuncture; Test type: Equivalence — a=0.05; p = 0.729, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | No Acupuncture/Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Acupuncture/Acupuncture (N=14)
Hospitalization (Cardiac disorders) | 2 (2) — Subjects were hospitalized for worsening heart failure, which was not unanticipated since a diagnosis of heart failure and a decreased left ventricular ejection fraction were required for study inclusion. Hospitalizations were subject-reported.

LIMITATIONS AND CAVEATS:
These results should be interpreted with caution. With only 10 subjects, the study may be under-powered to detect a significant difference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No